CLINICAL TRIAL: NCT02829554
Title: Differential Influences of Integral and Incidental Emotion on Cancer-Related Judgments and Decision Making
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916142; 16-C-N142
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Cancer; Overweight; Obesity
Keywords: Emotion; Judgment; Decision Making
MeSH Terms: conditions — Neoplasms; Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Respondents: US residents recruited to an on-line questionnaire through Amazon mTurk.

SUMMARY:
Background:

Researchers are testing new methods for research projects. They want to see how people respond to different types of communication, including videos. They also want to learn how people respond to life events and how they pay attention to computer tasks. They want to learn about how various risks and threats affect the way people make decisions.

Objectives:

To learn how different stimuli and events affect the way people make decisions.

Eligibility:

Adults ages 18 and older with a U.S. computer address

Design:

Participants will be recruited online.

Participants will take one of three studies online. Each study will take about a half hour.

Participants in Study 1 will watch a short video from a popular movie then answer questions. They will also complete 2 questionnaires. One will be about how likely they think it is that they will experience different risks and threats. The other will be about goals for behavior change.

Participants in Study 2 will write in detail about a life event. Then they will answer questions. They will also complete the same 2 questionnaires as Study 1.

Participants in Study 3 will pay close attention to words and images on a computer. They will answer questions about attitudes toward different behaviors, products, and experiences.

...

DETAILED DESCRIPTION:
Despite evidence that both integral (i.e., related to the decision) and incidental (i.e., unrelated to the decision) emotions influence cancer-related decision making, no research has systematically examined whether these two types of emotion generate similar patterns of influence, as predicted by decision-making models. This is important because incidental emotions are often used experimentally to draw causal conclusions about how emotions influence cancer-related decisions with the notion that results will generalize to produce knowledge about integral emotions as well. Across three studies, we plan to directly compare integral and incidental emotional influences on judgments and decisions related to cancer control. We plan to examine whether effects are contingent on the type of emotional influence (the discrete emotions anger and fear, or general positive affect) or type of emotion induction (video, autobiographical induction, or evaluative conditioning). Across experiments, we predict that emotion will influence both judgment and decision-making outcomes when the induced emotion is integral as well as when it is incidental. However, we predict that the magnitude of the effect of emotion on these types of responses will be significantly greater when emotions are integral to a judgment or decision, compared to when emotions are incidental.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults ages 18 and older with a U.S. computer address

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Studies 1a-3: general sample, nominally healthy individuals, recruited via Amazon mTurk, US residents only (age 18+) Study 2: three types of samples: 1) general sample, nominally healthy individuals, recruited via Amazon mTurk, US residents only (age 18+); 2) individuals who have been diagnosed with cancer (cancer survivors); 3) individuals who have low self-reported health
Sampling Method: Non-Probability Sample
Enrollment: 6242 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Risk perceptions | End of protocol
  Perceived susceptibility to cancer and other threats (self-report)
Intentions | End of protocol
  Intentions to engage in cancer and other threat-preventive behavior (self-report)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Ferrer, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States